CLINICAL TRIAL: NCT07117591
Title: Frequency of Restless Legs Syndrome and Its Impact on Sleep Quality in Patients With Pes Planus: A Multicenter Observational Study
Brief Title: Restless Legs Syndrome and Sleep Quality in Pes Planus
Acronym: FLAT-RLS
Status: Completed | Type: Observational
Sponsor: Bozok University (Other)
Collaborators: Ankara Etlik City Hospital (Other Government); Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gulseren Demir Karakilic, Assistant Professor, Principal Investigator, Bozok University
Other Study IDs: 2024/21
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Restless Legs Syndrome; Sleep Quality; Pain; Quality of Life; Pes Planus; Depression
Keywords: Pes Planus; Restless Legs Syndrome; Sleep Disturbance; Foot Pain; Anxiety; Depression; Quality of Life; Foot Function
MeSH Terms: conditions — Restless Legs Syndrome; Sleep Initiation and Maintenance Disorders; Pain; Flatfoot; Depression; Parasomnias; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: Participants in this group were clinically diagnosed with pes planus (flatfoot) by a physical medicine and rehabilitation specialist, based on physical examination findings. Individuals were aged between 18 and 65 years and presented with lower extremity pain. No intervention was applied. This group was evaluated using standardized questionnaires to assess the presence and severity of Restless Legs Syndrome, pain levels, emotional status, sleep quality, and quality of life.
- the Control group: This group included healthy volunteers between the ages of 18 and 65 who had no clinical signs of pes planus or lower extremity pain. Participants were matched to the patient group by age and sex. No medical or rehabilitative intervention was applied. They were evaluated using the same standardized tools to assess the presence of Restless Legs Syndrome, emotional status, sleep quality, and quality of life, for comparison with the patient group.

SUMMARY:
Pes planus, also known as flatfoot, is a common foot deformity that can affect the biomechanics of the lower limbs. However, its relationship with neurological conditions has not been studied extensively. Restless Legs Syndrome is a neurological disorder characterized by uncomfortable sensations in the legs and an urge to move them, especially during periods of rest, which can negatively affect sleep quality.

The aim of this multicenter cross-sectional study, conducted at Etlik Zübeyde Hanım Women's Health Training and Research Hospital, Etlik City Hospital in Ankara, and Yozgat City Hospital, is to determine the frequency of Restless Legs Syndrome in patients diagnosed with pes planus and to examine its effects on pain, emotional status, sleep quality, and quality of life. The study included 122 patients aged between 18 and 65 years with clinically diagnosed pes planus, and 120 healthy individuals matched for age and sex. Participants were assessed using the International Restless Legs Syndrome Study Group Diagnostic Criteria and Severity Rating Scale for Restless Legs Syndrome, the Visual Analog Scale and Foot Function Index for pain and foot function, the Hospital Anxiety and Depression Scale for emotional status, the Pittsburgh Sleep Quality Index for sleep quality, and the Short Form-36 Health Survey for quality of life.

DETAILED DESCRIPTION:
Pes planus, commonly known as flatfoot, is a frequent foot deformity characterized by a lowered medial longitudinal arch, which can affect lower limb biomechanics and overall posture. While its mechanical effects on the musculoskeletal system have been widely studied, the potential neurological and psychosocial implications of pes planus remain insufficiently explored.

Restless Legs Syndrome (RLS) is a neurological disorder marked by an uncontrollable urge to move the legs, often accompanied by unpleasant sensations. Symptoms typically worsen during rest or inactivity and can lead to significant sleep disturbances and reduced quality of life.

This multicenter cross-sectional observational study was designed to investigate the prevalence of RLS among patients clinically diagnosed with pes planus, and to evaluate the impact of RLS on pain severity, emotional well-being, sleep quality, and overall health-related quality of life.

The study was conducted between December 2024 and July 2025 at three tertiary care centers: Etlik Zübeyde Hanım Women's Health Training and Research Hospital, Etlik City Hospital in Ankara, and Yozgat City Hospital. A total of 242 participants were recruited, including 122 patients with clinically confirmed pes planus and 120 age- and sex-matched healthy controls without foot deformities or leg pain.

Inclusion criteria for patients were age between 18 and 65 years and a clinical diagnosis of pes planus by a physical medicine and rehabilitation specialist, based on physical examination. Exclusion criteria included the presence of systemic diseases such as diabetes mellitus, hypothyroidism, chronic renal failure, neuropathies, rheumatological conditions, history of foot surgery or fractures, and other conditions potentially affecting pain perception or neurological status.

Data collection included demographic information (age, sex, body mass index, educational status, smoking and alcohol use) and clinical variables (duration and severity of leg pain). The presence and severity of RLS were assessed using the International Restless Legs Syndrome Study Group Diagnostic Criteria and Severity Rating Scale, which are internationally recognized tools for diagnosis and quantification of symptom severity.

Pain intensity and foot function were measured using the Visual Analog Scale and the Foot Function Index, respectively. Emotional status was evaluated by the Hospital Anxiety and Depression Scale. Sleep quality was assessed with the Pittsburgh Sleep Quality Index, and overall quality of life was measured by the Short Form-36 Health Survey.

All assessments were performed by trained evaluators following a standardized protocol to ensure consistency across study sites. Data were collected through patient interviews, questionnaires, and clinical examinations.

The primary objective was to determine the frequency of Restless Legs Syndrome among pes planus patients compared to healthy controls. Secondary objectives included evaluating the relationship between RLS severity and pain intensity, emotional status, sleep quality, and quality of life.

This study aims to shed light on the complex interaction between biomechanical foot deformities and neurological symptoms, with the goal of informing comprehensive, multidisciplinary treatment approaches for patients with pes planus.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Clinical diagnosis of pes planus by a physical medicine and rehabilitation specialist (for patient group)
* Ability to understand and provide written informed consent
* For control group: healthy individuals matched by age and sex without pes planus or leg pain

Exclusion Criteria:

* History of diabetes mellitus, hypothyroidism, chronic renal failure, neuropathic disorders, vasculitis, lumbar disc disease
* Previous foot fracture or surgery
* Rheumatologic diseases affecting pain perception (e.g., rheumatoid arthritis, ankylosing spondylitis, fibromyalgia)
* Significant circulatory disorders in lower extremities
* Undergoing chemotherapy or radiotherapy
* Cognitive impairment preventing questionnaire completion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes adult patients aged 18-65 with clinically diagnosed pes planus and age- and sex-matched healthy controls without foot deformity or leg pain. Participants were recruited from three tertiary hospitals in Turkey and evaluated for Restless Legs Syndrome, pain, emotional status, sleep quality, and quality of life.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
The International Restless Legs Syndrome Study Group Diagnostic Criteria | At baseline
  Restless Legs Syndrome will be diagnosed using the International Restless Legs Syndrome Study Group Diagnostic Criteria, which consist of five essential clinical criteria. All criteria must be met for diagnosis. These include: (1) an urge to move the legs; (2) symptoms that begin or worsen during rest or inactivity; (3) symptoms relieved by movement; (4) symptoms worse in the evening or at night; and (5) symptoms not solely accounted for by another medical or behavioral condition.This tool, originally developed in 1995 and revised in 2014, includes five essential diagnostic criteria and is based solely on clinical history. All criteria must be met for a diagnosis of restless legs syndrome
The International Restless Legs Syndrome Study Group Criteria Severity Rating Scale | At baseline
  The severity of Restless Legs Syndrome symptoms will be assessed using the International Restless Legs Syndrome Study Group Severity Rating Scale. This is a validated 10-item questionnaire that evaluates symptom intensity, frequency, sleep disruption, and the psychosocial impact of Restless Legs Syndrome. Each item is scored from 0 to 4, with total scores ranging from 0 to 40. Severity is categorized as mild (1-10), moderate (11-20), severe (21-30), and very severe (31-40). The scale has been validated for use in Turkish populations.Total severity score (range 0-40) and severity category distribution (mild/moderate/severe/very severe).
The Pittsburg Sleep Quality Index | At baseline
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index, a 24-item self-reported questionnaire that evaluates sleep quality and disturbances over the past month. Scores range from 0 to 21, with higher scores indicating poorer sleep quality. A total score of 5 or above is used to define poor sleep quality. The index has been validated in Turkish populations.Total Pittsburgh Sleep Quality Index score and proportion of participants classified as poor sleepers (score ≥5)

SECONDARY OUTCOMES:
The Foot Function Index | At baseline
  Foot function will be evaluated using the Foot Function Index, a 23-item questionnaire assessing three subdomains: pain, disability, and activity limitation. Each item is scored on a scale to quantify the impact of foot problems on daily activities. The total score reflects overall foot function impairment, with higher scores indicating greater dysfunction. The Turkish version of this scale has been validated for reliability and validity.Total Foot Function Index score and scores of subdomains (pain, disability, activity limitation)
The Hospital Anxiety and Depression Scale | At baseline
  Anxiety and depression symptoms will be assessed using the Hospital Anxiety and Depression Scale, a 14-item self-report questionnaire consisting of two subscales: anxiety and depression. Each subscale includes 7 items scored to evaluate symptom severity. Scores of 8 or above on each subscale indicate clinically significant anxiety or depression. The scale has been validated in Turkish populations. Subscale scores for anxiety and depression; number and percentage of participants scoring 8 or above on each subscale
SF-36 | At baseline
  Quality of life will be measured using the Short Form-36 (SF-36) Health Survey, a 36-item self-administered questionnaire assessing eight health domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health. Each subscale is scored from 0 to 100, with higher scores indicating better perceived health status. The Turkish version of the SF-36 has been validated and is widely used in clinical research. Scores on each of the eight SF-36 subscales and composite physical and mental health scores

CONTACTS AND LOCATIONS:
Overall Officials: Gülseren Demir Karakılıç, Asst Prof, Principal Investigator — Yozgat Bozok University
Locations (1):
- Yozgat Bozok University Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) from this study, including de-identified demographic, clinical, and questionnaire data, will be available upon reasonable request after publication of the study results. Requests should be submitted to the corresponding author, who will evaluate the request for ethical and privacy compliance before sharing
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD and supporting documents will be available starting from the date of publication of the study results and will remain available for at least five years.
Access Criteria: Access to the IPD and supporting information will be granted to qualified researchers upon submission of a reasonable request explaining the research purpose. The corresponding author and ethics committee will review the requests to ensure compliance with ethical standards and protection of participant confidentiality. Data will be shared via secure data transfer methods after signing a data use agreement.

REFERENCES:
- [Background] Kocyigit H (1999) Turkish validity and reliability of short-form 36. Drug Treat 12:102-106
- [Background] Ağargün MY (1996) Validity and reliability of Turkish version of Pittsburgh Sleep Quality Index. Türk Psikiyatri Dergisi 7:107
- [Background] Aydemir O, Güvenir T, Küey L, Kültür S (1997) Reliability and validity of the Turkish version of hospital anxiety and depression scale. Turkish journal of psychiatry 8:280-287
- [Background] Ay E (2017) Huzursuz bacaklar sendromunda kullanılan uluslararası huzursuz bacaklar sendromu çalışma grubu şiddet ölçeğinin türkçe geçerlilik ve güvenilirliğinin araştırılması. In. Sağlık Bilimleri Enstitüsü.
- [Background] Allen RP, Picchietti DL, Garcia-Borreguero D, Ondo WG, Walters AS, Winkelman JW, Zucconi M, Ferri R, Trenkwalder C, Lee HB; International Restless Legs Syndrome Study Group. Restless legs syndrome/Willis-Ekbom disease diagnostic criteria: updated International Restless Legs Syndrome Study Group (IRLSSG) consensus criteria--history, rationale, description, and significance. Sleep Med. 2014 Aug;15(8):860-73. doi: 10.1016/j.sleep.2014.03.025. Epub 2014 May 17. PMID 25023924
- [Background] YALIMAN A, ŞEN Eİ, ESKİYURT N, BUDIMAN-MAK E (2014) Ayak Fonksiyon İndeksi'nin Plantar Fasiitli Hastalarda Türkçe'ye Çeviri ve Adaptasyonu. Turkish Jour